CLINICAL TRIAL: NCT05501873
Title: Real World Data Collection in Subjects Treated With the FARAPULSE Pulsed Field Ablation System
Acronym: FARADISE
Status: Active, not recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PF114
Record Dates: First submitted 2022-08-12; First posted 2022-08-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: FARAPULSE Pulsed Field Ablation system — Any subject who has signed the informed consent and for whom the FARAPULSE Pulsed Field Ablation system has been inserted into the body, and pulsed field ablation treatment has been received, are assigned to the treatment group.

SUMMARY:
The goal of any novel design or therapeutic strategy to treat atrial fibrillation is to restore normal sinus rhythm and to reduce or eliminate the symptoms due to rapid atrial response.

Boston Scientific has developed the FARAPULSE™ Pulsed Field Ablation therapy that uses irreversible electroporation to induce cell death.

This Registry is intended to obtain purely observational and prospective real world data and to provide continued evidence on the safety and effectiveness when the FARAPULSE™ pulsed field ablation System is used per hospitals' standard of care.

DETAILED DESCRIPTION:
This Registry is intended to obtain purely observational and prospective real world data about the cardiac ablation procedure in subjects treated with the FARAPULSE™ Pulsed Field Ablation system, to provide continued evidence on the safety and effectiveness of the FARAPULSE™ Pulsed Field Ablation (PFA) System when used per hospitals' standard of care, and to learn the effect of the Pulsed Field Ablation treatment on Quality Of Life in a real-world setting. The study will enroll approximately 1000 to 1500 subjects, in up to 100 sites in Europe (with the potential for expansion of the study to Middle East, Africa and/or Asia Pacific).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects intended to be treated with the FARAPULSE™ Pulsed Field Ablation system for cardiac tissue ablation, per physician's medical judgement, and as per hospitals' standard of care
2. Subjects who are willing and capable of providing informed consent
3. Subjects who are willing and capable of participating in all testing associated with this clinical study at an approved clinical investigational center
4. Subjects whose age is 18 years or above, or who are of legal age to give informed consent specific to state and national law

Exclusion Criteria:

1. Subjects with a current interatrial baffle or patch
2. Subjects with a known or suspected atrial myxoma
3. Subjects with a myocardial infarction within 14 days prior to enrollment
4. Subjects with a recent (within 30 days prior to enrollment) Cerebral Vascular Accident (CVA)
5. Subjects who do not tolerate anticoagulation therapy
6. Subjects with an active systemic infection *
7. Subjects with a presence of atrial known thrombus *
8. Subjects with a known inability to obtain vascular access
9. Subjects who are pregnant or planning to be pregnant
10. Subjects with atrial fibrillation that is secondary to electrolyte imbalance, thyroid disease, alcohol, or other reversible / non-cardiac causes
11. Subjects with any prosthetic heart valve, ring or repair including balloon aortic valvuloplasty
12. Subjects with a contraindication to an invasive electrophysiology procedure where insertion or manipulation of a catheter in the cardiac chambers is deemed unsafe per physician's medical judgement, such as, but not limited to, a recent previous cardiac surgery (eg. ventriculotomy or atriotomy, CABG, PTCA/PCI/coronary stent procedure/unstable angina) and/or in patients with congenital heart disease where the underlying abnormality increases the risk of the ablation (e.g., severe rotational anomalies of the heart or great vessels)
13. Subjects with a life expectancy of ≤ 1 year per investigator's opinion
14. Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments. Each instance must be brought to the attention of the sponsor to determine eligibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects enrolled in the FARADISE study will be clinically indicated for an ablation procedure with the FARAPULSE™ Pulsed Field Ablation system, per physician's medical judgement, and according to the hospitals' standard of care
Sampling Method: Probability Sample
Enrollment: 1173 (Actual)
Dates: Start 2023-03-24 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | 12 monhts
  Failure-free rate at 12 months post index procedure

SECONDARY OUTCOMES:
Safety endpoint | 12 months
  Composite of device- or procedure-related serious adverse events at early onset or chronic onset

CONTACTS AND LOCATIONS:
Locations (48):
- Australia (3):
  - Prince Charles Hospital, Brisbane
  - Fiona Stanley Hospital, Murdoch
  - John Hunter Hospital, Newcastle
- Allgemeines Krankenhaus AKH, Vienna, Austria
- Belgium (3):
  - AZ Sint Jan Hospital, Bruges
  - Hartcentrum Hasselt Jessa Ziekenhuis Campus Virga Jesse, Hasselt
  - CHR de la Citadelle, Liège
- Czechia (2):
  - Neuron Medical in Brno, Brno
  - Nemocnice Ceske Budejovice a.s., České Budějovice
- Tays Heart Hospital, Tampere, Finland
- France (6):
  - CHU Grenoble, Grenoble
  - Hopital Saint Philibert-Hospital, Lomme
  - Hopital Prive du Confluent SAS, Nantes
  - Clinique Ambroise Pare-Hospital, Neuilly
  - Centre Cardiologique du Nord, Saint-Denis
  - Clinique Pasteur Toulouse, Toulouse
- Germany (7):
  - Universitaetsklinikum Aachen (UKA), Aachen
  - Facharztzentrum Dresden-Neustadt Betriebsgesellschaft mbH, Dresden
  - Georg-August-Universitaet Goettingen, Göttingen
  - St Georg Asklepios, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Staedisches Klinikum Karlsruhe, Karlsruhe
  - University Hospital of Muenster, Münster
- Greece (2):
  - Henry Dunant hospital, Athens
  - Onassis Cardiac Surgery Center, Athens
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Semmelweis University, Budapest, Hungary
- Mater Private Hospital, Dublin, Ireland
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Italy (5):
  - Az. Osp. Lancisi-Hospital, Ancona
  - Casa Di Cura 'Montevergine' S.P.A., Mercogliano
  - Ospedale Rivoli, Rivoli
  - Ospedale Isola Tiberina Gemelli Isola, Roma
  - Ospedale San Bortolo de Vicenza, Vicenza
- Institut Jantung Negara, Kuala Lumpur, Malaysia
- Princesse Grace, Monaco, Monaco
- Netherlands (2):
  - Catharina Ziekenhuis, Eindhoven
  - St. Antonius Ziekenhuis, Nieuwegein
- Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego, Warsaw, Poland
- Hospital de Santa Cruz, Carnaxide, Portugal
- King Fahd Armed Forces Hospital, Jeddah, Saudi Arabia
- Spain (4):
  - Centro Especial Ramon y Cajal, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario La Fe, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- United Kingdom (2):
  - Royal Papworth Hospital, Cambridge
  - Liverpool Heart & Chest Hospital, Liverpool

IPD SHARING:
Plan to Share IPD: No